CLINICAL TRIAL: NCT02018081
Title: Population Pharmacokinetics of Levofloxacin in Intensive Care Patients With Severe Community-acquired Pneumonia.
Brief Title: Pharmacokinetics of Levofloxacin in Intensive Care Unit
Acronym: LEVO-PHARM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10 150 02
Record Dates: First submitted 2013-07-04; First posted 2013-12-23 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Intensive Care Unit Syndrome; Community-acquired Pneumonia
Keywords: pharmacokinetic study : open, prospective, monocentric
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Levofloxacin; Pharmacogenomic Variants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levofloxacin (Experimental): Population having a community-acquired pneumonia of which the indication of the treatment is administration of Levofloxacin
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin — 8 blood sampling by patients between the 48th and 60th
  Other Names: pharmacokinetic

SUMMARY:
The aim of this study is 1. to describe levofloxacin pharmacokinetics in ICU patients suffering from pneumonia with taking into account physio-pathological parameters. 2. to verify clinical and bacteriological efficiency and to know if the peak/Minimum Inhibitory Concentration (MIC) ratio > 5 and Area Under Curve (AUC) /Minimum Inhibitory Concentration(MIC) ratio > 125. No therapeutic drug monitoring will be performed in this study.

ELIGIBILITY:
Inclusion Criteria:

* severe community-acquired pneumonia due to a strain sensible to levofloxacin
* Age > 18 years
* Informed consent
* SAPS II (simplified acute physiological score) > 20 Awaited duration of survival higher than 7 days

Exclusion Criteria:

* Historic of allergy to levofloxacin
* Resistant strain to levofloxacin
* Pregnancy
* Contra-indications of levofloxacin use, renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Levofloxacin dosage regimen, time of administration and time of blood sampling, levofloxacin serum concentrations. | Levofloxacin concentration assessment at 8 different time points during 12h

SECONDARY OUTCOMES:
Efficiency (clinical,bacteriological, pharmacodynamic) | 12 hours
  age, weight, height, sex, SAPS II, blood urea nitrogen (BUN), creatinine, mechanical ventilation, leukocytes, haemoglobin, procalcitonin, creatinine clearance, proteins, MIC of the strain.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard GEORGES, MD, PhD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France